CLINICAL TRIAL: NCT01562522
Title: Evaluation of the Effect of Psycho-oncological Intervention on Well-being of Patients With Advanced Prostate Cancer on LHRH Analogs and Their Partners. A Randomized Controlled Pilot Study.
Acronym: EXPEDIENT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrolment; only 6 subjects enrolled and they were all screen failures.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A-95-52014-192; 2011-004819-24 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-26 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Psychological counseling
- Control group (No Intervention)

INTERVENTIONS:
Other: Psychological counseling — Attendance at 7 group sessions, consisting of 5-6 couples, preceded by an intake consultation. Total intervention time: 16 weeks.
  Arms: Intervention group

SUMMARY:
The purpose of the protocol, is to assess the feasibility of conducting a larger trial to evaluate the effect of a psychological intervention on the well-being of patients on luteinizing hormone-releasing hormone (LHRH) analogs in the treatment of prostate cancer and their partners.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer on biopsy
* Locally advanced or metastasised prostate cancer in need of hormonal treatment.
* On LHRH analogue treatment for a minimum of 5 months (at inclusion)
* Having a female partner
* Patients and their partner are able to fill out questionnaires, attend group sessions and give consent

Exclusion Criteria:

* Serious psychiatric difficulties
* Life expectancy < 12 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Sufficient interest in participation | Up to the end of 16 weeks of the intervention period
  Determined by achievement of all of the following:
  * Number of participants (couples) recruited in 18 months in the participating centres. Achieved by recruitment of 50 couples.
  * Number of participants (couples) informed personally about the study consent to participate. To be achieved by 20% of couples.
  * Number of participants in group 1 that attend at least 70% of the sessions. To be achieved by 80% of participants.
Preliminary improvement in well-being | After the intervention period of 16 weeks
  Improved - Group 1 improve more than group 2 on at least one of the outcome measures (includes HADS, EORTC QLQ-C30 or Maudsley Marital Questionnaire).
  Worsened - Group 1 should not worsen more than group 2 on any of the outcome measures.

SECONDARY OUTCOMES:
Change in quality of life questionnaire QLQ-C30 scores | Baseline (T0), after the intervention period of 16 weeks (T1) and 1 year (T2)
Change in quality of life questionnaire QLQ-PR25 scores | Baseline(T0), after the intervention period of 16 weeks (T1) and 1 year (T2)
Difference in relationship satisfaction (Maudsley Marital Questionnaire) | Baseline (T0), after the intervention period of 16 weeks (T1) and 1 year (T2)
Difference between level of depression and anxiety (HADS) | Baseline (T0) and 1 year (T2)
Change in Hospital Anxiety and Depression Scale (HADS) scores | Baseline (T0), after the intervention period of 16 weeks (T1)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Oncology, Study Director — Ipsen
Locations (3):
- Netherlands (3):
  - St. Antonius Hospital, Nieuwegein
  - Diakonessenhuis, Utrecht
  - Zuwe Hofpoort Ziekenhuis Woerden, Netherlands, Woerden